CLINICAL TRIAL: NCT05952102
Title: Role of Nigella Sativa Oil as an Adjuvant Therapy in the Treatment of Pediatric Pneumonia
Brief Title: Nigella Sativa as an Adjuvant Therapy in the Treatment of Pediatric Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Zaki Elmeazawy (Other)
Responsible Party: Sponsor-Investigator, Rehab Zaki Elmeazawy, Doctor, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nigella Sativa in Pneumonia
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Nigella Sativa Oil as an Adjuvant Therapy in the Treatment of Pneumonia
Keywords: Nigella Sativa Oil; Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 52 children with community acquired pneumonia will receive Nigella sativa oil capsules (Experimental): 52 children with community-acquired pneumonia will receive Nigella sativa oil in capsules at a dose of 40 mg/kg/day (8), as an adjunct therapy to the usual pneumonia treatment till the recovery of the disease.
  Interventions: Drug: Nigella Sativa Oil capsule
- 52 children (No Intervention): 52 children with community-acquired pneumonia with the usual pneumonia treatment as a control group

INTERVENTIONS:
Drug: Nigella Sativa Oil capsule — Nigella Sativa Oil as an Adjuvant Therapy in the Treatment of Pediatric Pneumonia
  Other Names: Black seed oil capsule
  Arms: 52 children with community acquired pneumonia will receive Nigella sativa oil capsules

SUMMARY:
Nigella sativa is the world's oldest immunomodulator. The main active component in Nigella sativa is thymoquinone. Research shows thymoquinone has antioxidant, anti-inflammatory, and antimicrobial effects. Based on these observations on the pharmacological activities of Nigella sativa, the potential therapeutic efficacy of N. Sativa was proposed in CAP.

DETAILED DESCRIPTION:
The aim of this work is to assess the benefit of oral Nigella Sativa oil supplementation, in addition to standard antibiotic and other supportive therapy, in the management of hospitalized children with pneumonia admitted to the Pulmonology Unit, Pediatric Department.

Primary outcome:

1- The duration of clinical manifestations of pneumonia including time taken for normalization of respiratory rate, temperature, and oxygen.

saturation, chest in drawing, hypoxia, lethargy, and inability to feed 2- The duration of hospital stay.

Secondary outcome:

1. Discharge or death of the patient.
2. Occurrence of pneumonia complications.

ELIGIBILITY:
Inclusion Criteria:

* Signs and symptoms of lower respiratory tract infections (LRTI) (LRTI was defined as ≥ 1 of the following: new or different cough or sputum production, chest pain, dyspnea, tachypnea, or abnormal auscultatory findings).
* Focal findings on chest x-ray indicating pneumonia.

Exclusion Criteria:

* Children with immunodeficiency, chronic lung disease, malignancy, congenital lung anomalies, underlying disorder impacting respiration i.e. genetic, metabolic, neuromuscular disorders….etc, children with CHD affecting the pulmonary blood flow

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | 3 days
  Time taken for normalization of respiratory rate
Temperature | 3 days
  Duration of defeverness
Oxygen saturation | 3 days
  Duration of normal oxygen saturation
Feeding | 3 days
  Duration of improvement of feeding
Respiratory distress | 7 days
  Duration of improvement of respiratory distress
Hospital stays | 14 days
  Duration of hospital stay

SECONDARY OUTCOMES:
Mortality | 30 days
  Discharge or death of the patient
Pneumonia complications | 30 days
  Occurrence of pneumonia complications

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa E. Fayed, MBBS, Study Chair — Tanta University
Locations (1):
- Faculty of Medicine, Tanta, Gharbia Governorate, Egypt